CLINICAL TRIAL: NCT03535090
Title: High-dose Intravenous Methylprednisolone Therapy in Patients With Graves' Orbitopathy is Associated With the Increased Activity of Factor VIII
Brief Title: Coagulation After Intravenous Methylprednisolone Administration
Status: Completed | Type: Observational
Sponsor: Piotr Miskiewicz (Other)
Responsible Party: Sponsor-Investigator, Piotr Miskiewicz, MD, PhD, Medical University of Warsaw
Organization: Medical University of Warsaw (Other)
Other Study IDs: IVMPCoagulation
Record Dates: First submitted 2018-04-29; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Graves' Disease; Graves Ophthalmopathy; Blood Coagulation; Venous Thromboembolism
Keywords: Graves' Disease; Graves Ophthalmopathy; Blood Coagulation; Venous Thromboembolism; Methylprednisolone
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy; Thrombosis; Venous Thromboembolism | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood was collected in the morning following a 12 hour fast. This was utilized for preparation of serum, 3.2% sodium citrate plasma, and citrate platelet - poor plasma after double centrifugation. Hemostatic parameters were analyzed within 1 - 1.5 hour after blood sampling, except for FVIII activity measured in platelet - poor plasma stored frozen at -70°C until assay.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- active, moderate-to-severe GO: Each participant received IVMP according to EUGOGO recommendations (cumulative dose of methylprednisolone 4.5 g, treatment duration 12 weeks in single weekly intravenous pulses, first 6 weeks 0.5g of IVMP, next 6 weeks 0.25g of IVMP).
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone

SUMMARY:
The alterations of coagulation and fibrinolysis parameters have been described in patients with endogenous Cushing's syndrome (CS) and those treated with glucocorticosteroids (GCs). The change in hemostatic process is associated with an increased risk of venous thromboembolic events (VTE) and pulmonary embolism (PE). Anticoagulation prophylaxis reduces thromboembolic complications in endogenous and exogenous hypercortisolism. The impact of the intravenous GCs therapy on hypercoagulability, however, remains unclear and perplexing. According to the European Group On Graves' Orbitopathy (EUGOGO), patients with active, severely symptomatic and sight-threatening Graves' orbitopathy (GO) should be treated with high dose intravenous methylprednisolone (IVMP) pulses. There are, however, reports of fatal side effects that may be associated with this therapy (e.g.: PE, myocardial infarction, severe cerebrovascular events, acute liver damage and sudden death). For this reason, the cumulative dose of IVMP should not exceed 8 g within each treatment course, and pulses should not be given on consecutive or alternate days, except for the case of dysthyroid optic neuropathy. Nevertheless, even smaller cumulative therapy may be associated with fatal cardiovascular complications. Hence the aim of our study was to evaluate the effects of IVMP therapy on hemostatic process in patients with GO. All of patients were treated according to EUGOGO recommendations with standard doses of methylprednisolone with standard recommended schedule. Inclusion criterion for the therapy was according to EUGOGO guidelines moderate-to-severe and active GO (12 pulses of IVMP 6x0.5g followed by 6x0.25g every week).

DETAILED DESCRIPTION:
The end point of the study was a change in hemostatic variables' levels in laboratory tests. There were short- and long-term hemostatic changes analysed during IVMP therapy: comparisons of laboratory tests before, 24h and 48h after selected pulses, and between the beginning of 1st, 6th and 12th IVMP pulses, respectively. Hemostatic variables that were evaluated: factor [F] II, FV, FVII, FVIII, fibrinogen, antithrombin, activated partial thromboplastin time, prothrombin time, platelets and D - dimer. Moreover, analyses were performed concerning clinical data (such as age, sex, body mass index, smoking, duration time of GO, presence of hypertension, basal markers of thyroid function) between independent groups (patients with initially increased/reduced selected markers versus without increased/reduced selected markers).

ELIGIBILITY:
Inclusion Criteria:

* active, moderate-to-severe Graves' orbitopathy according to EUGOGO classification
* euthyroidism for at least 1 month
* completion of at least first six IVMP pulses

Exclusion Criteria:

* medical history of thromboembolic events
* cardiovascular morbidity (chronic heart failure, cardiovascular heart disease)
* uncontrolled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg)
* liver disease (>3x increase of alanine aminotransferase and/or aspartate aminotransferase)
* active inflammation
* nephritic syndrome
* active neoplastic disease
* previous GCs therapy within the last 6 months
* trauma/surgery within the last 3 months
* pregnancy or a bedridden state
* use of: heparin, vitamin K antagonists, antiplatelet drugs, contraceptives or hormone replacement therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Endocrine Department
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Change in activity of coagulation factor VIII from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in activity of coagulation factor VIII from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in of activated partial thromboplastin time (seconds) from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in activated partial thromboplastin time (seconds) from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks

SECONDARY OUTCOMES:
Change in activity of coagulation factor II from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in activity of coagulation factor V from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in activity of coagulation factor VII from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in prothrombin time (seconds) from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in fibrinogen (mg/dl) from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in D-Dimer (ng/dl) from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in PLT count from baseline (before administration of methylprednisolone) to 24 hours after first intravenous pulse | 24 hours
Change in activity of coagulation factor II from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in activity of coagulation factor V from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in activity of coagulation factor VII from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in prothrombin time (seconds) from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in fibrinogen (mg/dl) from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in D-Dimer (ng/dl) from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks
Change in PLT count from baseline (before therapy) to the end of the course of therapy with methylprednisolone | 12 weeks

OTHER OUTCOMES:
Change in activity of coagulation factor VIII from baseline (before administration of methylprednisolone) to 48 hours after the first intravenous pulse | 48 hours
Change of activated partial thromboplastin time (seconds) from baseline (before administration of methylprednisolone) to 48 hours after the first intravenous pulse | 48 hours
Change in activity of coagulation factor VIII from baseline (before therapy) to the sixth pulse of the methylprednisolone | 6 weeks
Change activated partial thromboplastin time (seconds) from baseline (before therapy) to the sixth pulse of the methylprednisolone | 6 weeks

IPD SHARING:
Plan to Share IPD: Yes
The collected data will be shared in a publication. It includes all laboratory results from all points of evaluation: hemostatic variables- factor [F] II, FV, FVII, FVIII, fibrinogen, activated partial thromboplastin time, prothrombin time, international normalized ratio of prothrombin time, platelet count and D - dimer.
Supporting Information: Study Protocol, SAP
Time Frame: The results of the study will be published in 2018